CLINICAL TRIAL: NCT07220889
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Single and Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MDI-2517 in Healthy Participants
Brief Title: Single Ascending Dose and Multiple Ascending Dose Evaluation of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MDI-2517 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MDI Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDI-2517-01-002
Record Dates: First submitted 2025-10-19; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Safety After Oral Intake
Keywords: single ascending dose; multiple ascending dose; safety; pharmacokinetics; pharmacodynamics; MDI-2517

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- SAD 1 (Active Comparator): SAD cohort 1 will receive a single oral dose of 2400 mg of MDI-2517 or matching placebo
  Interventions: Other: Placebo; Drug: MDI-2517 2400mg
- SAD 2 (Active Comparator): SAD cohort 2 will receive a single oral dose up to 3600 mg of MDI-2517 or matching placebo.
  Interventions: Other: Placebo; Drug: MDI-2517 3600mg
- MAD 1 (Active Comparator): MAD cohort 1 will receive a total daily dose of 800 mg of MDI-2517 or matching placebo administered either once daily (QD) or twice daily (BID).
  Interventions: Drug: MDI-2517 800mg; Other: Placebo
- MAD 2 (Active Comparator): MAD cohort 2 will receive a total daily dose of up to 1600 mg of MDI-2517 or matching placebo administered either QD or BID.
  Interventions: Other: Placebo; Drug: MDI-2517 1600mg
- MAD 3 (Active Comparator): MAD cohort 3 will receive a total daily dose of up to 2400 mg of MDI-2517 or matching placebo administered either QD or BID.
  Interventions: Other: Placebo; Drug: MDI-2517 2400mg

INTERVENTIONS:
Drug: MDI-2517 800mg — 800mg MDI-2517 will be administered
  Arms: MAD 1
Other: Placebo — Matching Placebo
Drug: MDI-2517 1600mg — MDI-2517 1600mg will be adminstered
  Arms: MAD 2
Drug: MDI-2517 2400mg — MDI-2517 2400mg will be administered
  Arms: MAD 3; SAD 1
Drug: MDI-2517 3600mg — MDI-2517 3600mg will be administered
  Arms: SAD 2

SUMMARY:
The goal of this clinical trial is to learn if drug MDI2517 is safe and to learn more about its drug effects in healthy participants. Healthy participants will take single or multiple doses of drug and the safety and drug levels will be measured.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if drug MDI2517 is safe and to learn more about its drug effects in healthy participants. Healthy participants will take single or multiple doses of drug and the safety and drug levels will be measured. Healthy participants will be monitored for adverse events, laboratory test changes, changes in vital signs, electrocardiogram and the plasma drug levels will be measured. The amount of the drug and its metabolites in urine and blood will be measured. Blood and urine will be used to evaluate the effects of MDI-2517.

ELIGIBILITY:
Inclusion Criteria:

1. Capable to understand the study procedures and providing signed informed consent as described Section 8.2, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Healthy male and female participants 18 to 55 years of age inclusive, at the time of signing the informed consent.
3. Body weight of a minimum 50 kg for men and 45 kg for women and body mass index (BMI) within the range of 18.5 to 32 kg/m2
4. Participants who are generally healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring.
5. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Female participants should be of nonchildbearing potential (postmenopausal i.e., spontaneous amenorrhea for at least 12 months prior to dosing with confirmatory follicle-stimulating hormone [FSH] > 40 mIU/mL, or premenopausal and surgically sterilized), or of childbearing potential who agree to take highly effective contraceptive measures throughout the trial (see Section 11.15 for highly effective contraceptive guidance). Sexually active female participants of childbearing potential with non-sterile male partners, and sexually active non-surgically sterile male participants with female partners of childbearing potential will be required to use highly effective double contraceptive method. Women of childbearing potential and those with less than 24 weeks from menopause must undergo a urine pregnancy test at screening and result must be negative.
6. Ability to refrain from consumption of Seville oranges, grapefruit or grapefruit juice, pomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices from 7 days before participants check into the clinical site until collection of the final PK sample for each participant.
7. Ability to abstain from ingesting caffeine- or xanthine-containing products (eg, coffee, black/green tea, cola drinks, and chocolate) or energy drinks for 48 hours before participants check into the clinical site until after collection of the final PK and/or PD sample.
8. Ability to abstain from alcohol for 24 hours before admission to the clinical site until after collection of the final PK and/or PD sample.
9. Ability to swallow multiple tablets within a 10 minute window.

Exclusion Criteria:

1. Major medical illness or unstable medical condition within 6 months of screening that in the opinion of the investigator may interfere with the participant's ability to comply with study procedures and abide by study restrictions, or with the ability to interpret safety data that would prevent completion of study procedures or assessments.
2. Any clinically significant abnormal finding at Screening during the physical examination or a clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Chronic or ongoing active infectious disease requiring systemic treatment including, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, and tuberculosis.
4. Any acute infections within 14 days of screening.
5. Live attenuated vaccines received within 1 month of screening. Other vaccines, including coronavirus 2019 (COVID-19) vaccine, within 14 days prior to Screening.
6. Participants known or suspected of not being able to comply with this study protocol (eg, due to alcoholism, drug dependency or psychological disorder)
7. Laboratory values as follows:

   1. Any clinically significant lab abnormalities
   2. AST or ALT; > the upper limit of normal (ULN)
   3. Total bilirubin > 1.5 times ULN (isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin is < 35%)
   4. Platelet counts < 150 × 109/L or > 450 × 109/L
   5. Hemoglobin outside of normal limits
   6. Coagulation tests (prothrombin time, partial thromboplastin time) outside of normal limits
8. Screening corrected QT interval (QTc) > 450 milliseconds for males and > 470 ms for females. The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF), machine read or manually overread.
9. Screening estimated glomerular filtration rate (eGFR) using 2021 CKD-EPI method <90 mL/min/1.73m2
10. Positive serology test results for Hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen and antibody at screening. Positive evaluation for COVID-19 infection.
11. History of significant allergic reactions (eg, anaphylactic reaction, hypersensitivity, angioedema) to any drug.
12. Use of prescription or nonprescription drugs, including vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication through the final study visit, unless in the opinion of the investigator and Medical Monitor the medication will not interfere with the study procedures or compromise participant safety with the exception of oral contraception or the occasional use of acetaminophen (up to 2 g daily). Use of monoamine oxidase inhibitors and St. John's Wort within 30 days of dosing.
13. Treatment with nonsteroidal anti-inflammatory drugs (NSAIDs, eg, acetylsalicylic acid) or selective serotonin reuptake inhibitors within 7 days prior to screening through the final study visit.
14. Use of tobacco products or uses other nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, inhalers or vapes) from 3 months before screening until final follow-up visit. Use of cigarettes 3 months before screening until final visit.
15. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 7 units for women or 14 units for men of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%) through the final study visit.
16. History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening through the final study visit.
17. History of hypersensitivity to platelet concentrates or human plasma proteins.
18. Any type of known platelet function disorder.
19. Individuals with increased risk of thrombotic events (eg, history of pulmonary embolism or thrombosis).
20. Any blood product donation given or received within 3 weeks of screening or loss of 500 mL or more of whole blood within 8 weeks prior to dosing.
21. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration. Previously received MDI-2517 study drug or placebo in this study.
22. Positive pregnancy test or lactating female participant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-11-04 (Estimated); Primary Completion 2026-05-04 (Estimated); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of single and multiple ascending oral doses of MDI-2517 in healthy participants | SAD cohorts are up to 34 days - up to 28 days for screening, 1 day of dosing (for SAD cohorts) and 6 days of monitoring. MAD cohorts are up to 40 days - up to 28 days for screening. 7 days of dosing (for MAD cohorts) 12 days of monitoring.
  Evaluate the safety of single and multiple ascending oral doses of MDI-2517 in healthy participants.
  This outcome will be measured using:
  the number of participants with adverse events (AEs), with abnormal laboratory tests results (chemistry, hematology, coagulation), abnormal vital signs and changes in electrocardiogram"
  * The type, incidence, severity, seriousness, and relatedness of adverse events (AEs)
  * The type, incidence, and severity of laboratory abnormalities and changes (chemistry, hematology, coagulation)
  * Changes in vital signs, and changes in electrocardiogram (ECG QT prolongation) at specified timepoints

SECONDARY OUTCOMES:
Evaluate the plasma pharmacokinetic (PK) profile of MDI-2517 following ascending single oral doses of MDI2517 in healthy participants | SAD cohorts are up to 34 days- Screening up to 28 days. 1 day of dosing (for SAD cohorts) and 6 days of monitoring.
  Evaluate the plasma pharmacokinetic (PK) profile of MDI-2517 following ascending single oral doses of MDI2517 in healthy participants. This outcome - the PK profile of MDI-2517- will be measured by analyzing blood samples measuring: Cmax; tmax; AUC0-24; AUC0-t; AUC0-inf; t½; λz; CL/F; Vz/F; and linearity factor)
Evaluate the plasma PK profile of MDI-2517 following ascending multiple oral doses of MDI-2517 in healthy participants | MAD cohorts are up to 40 days. Screening up to 28 days. dosing on days 1 to 7 (for MAD cohorts) and 12 days of monitoring.
  Evaluate the plasma PK profile of MDI-2517 following ascending multiple oral doses of MDI-2517 in healthy participants. This outcome - the PK profile of MDI-2517- will be measured by analyzing blood samples- and will be measured using: Cmax; Cmin; tmax; AUC0-24; AUC0-t; AUC0-inf (Day 1 only); t½; λz; CL/F; Vz/F; linearity factor; and accumulation index ratios for Cmax and AUCs.

OTHER OUTCOMES:
Determine the renal excretion of MDI-2517 and analysis of MDI-2517 and metabolites following multiple oral doses. | MAD cohorts are up to 40 days. Screening up to 28 days, dosing days 1-7 (for MAD cohorts) and 12 days of monitoring.
  Determine the renal excretion of MDI-2517 and possible analysis of MDI-2517 and metabolites following multiple oral doses. This outcome will be measured by: Analyzing concentrations of MDI-2517 in urine, Ae0-last: cumulative urinary excretion, percentage of dose excreted unchanged in urine • ClR: Renal clearance, calculated as Ae0-last /AUC 0-t)
Evaluate target engagement and pharmacodynamic (PD) effects of MDI-2517 following multiple oral doses | MAD cohorts are up to 40 days. Screening up to 28 days. Dosing days 1 to 7 (for MAD cohorts) and 12 days of monitoring.
  Evaluate target engagement and pharmacodynamic (PD) effects of MDI-2517 following multiple oral doses. This outcome - target engagement and the pharmacodynamic (PD) effects will be measured using: Blood, urine, and peripheral blood mononuclear cell (PBMC) collections to evaluate possible drug effects of MDI-2517. i.e. how the drug MDI-2517 effects the patient's blood and urine.

CONTACTS AND LOCATIONS:
Overall Officials: David Wyatt, MD, Principal Investigator — MDI Therapeutics, Inc.
Locations (1):
- 1951 NW 7th Avenue, Suite 180, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No